CLINICAL TRIAL: NCT04448340
Title: A Novel Machine Learning Algorithm to Predict the Lewy Body Dementias Using Clinical and Neuropsychological Scores
Brief Title: A Novel Machine Learning Algorithm to Predict the Lewy Body Dementias
Acronym: MLDLB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Anastasia Bougea, DR, National and Kapodistrian University of Athens
Other Study IDs: 251ATHENS HOSPITAL
Record Dates: First submitted 2020-06-21; First posted 2020-06-25 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Disease Dementia: the PDD group comprised of 58 patients fulfilling the Criteria for probable PDD of the Movement Disorders Society
  Interventions: Diagnostic Test: machine learning model
- Dementia with Lewy Bodies: the DLB group comprised of 40 patients, according to the recent revised criteria for probable DLB
  Interventions: Diagnostic Test: machine learning model

INTERVENTIONS:
Diagnostic Test: machine learning model — Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), were investigated for their ability to predict successfully whether patients suffered from PDD or DLB.

SUMMARY:
Parkinson's disease dementia (PDD) and Dementia with lewy bodies (DLB) are dementia syndromes that overlap in many clinical features, making their diagnosis difficult in clinical practice, particularly in advanced stages. We propose a machine learning algorithm, based only on non-invasively and easily in-the-clinic collectable predictors, to identify these disorders with a high prognostic performance.

DETAILED DESCRIPTION:
The algorithm will be develop using dataset from two specialized memory centers, employing a sample of PDD and DLB subjects whose diagnostic follow-up is available for at least 3 years after the baseline assessment. A restricted set of information regarding clinico- demographic characteristics, 6 neuropsychological tests (mini mental, PD Cognitive Rating Scale, Brief Visuospatial Memory test, Symbol digit written, Wechsler adult intelligence scale, trail making A and B) was used as predictors. Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), will be investigated for their ability to predict successfully whether patients suffered from PDD or DLB.

ELIGIBILITY:
Inclusion Criteria:

the PDD group comprised of patients fulfilling the Criteria for probable PDD of the Movement Disorders Society (b) the DLB group comprised of patients, according to the recent revised criteria for probable DLB .

Exclusion Criteria:

* major psychiatrics disorders, depression

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the PDD group comprised of patients fulfilling the Criteria for probable PDD and the DLB group.Patients will be enrolled from the register-based database of two clinics. The following data were collected: gender, age, education, hand dominance, Disease duration (years) and levodopa equivalent daily dose (LEDD). The burden of disease will be assess by the Movement Disorders Society-United Parkinson's Disease Rating Scale (MDS-UPDRS) part III in the Off medication state and the following six cognitive/behavioral tests: Mini-Mental State Examination (MMSE), PD- Cognitive Rating Scale (PD-CRS), Brief Visuospatial Memory test (BVMT-TR), Symbol digit written (SDMT), Trail making test (TMT A,B), Wechsler adultintelligence scale (WAIS-V). All patients will undergo brain MRI and blood test to exclude secondarycauses of dementia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
MMSE predictive for dlb or PDD | 1 year
  Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), will combine these tests in order to investigate for their ability to predict successfully whether patients suffered from PDD or DLB.
Parkinson's Disease - Cognitive Rating Scale (PD-CRS) predictive for DLB or PDD | 1 year
  Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), will combine these tests in order to investigate for their ability to predict successfully whether patients suffered from PDD or DLB.
Brief Visuospatial Memory Test (BVMT-TR) predictive for DLB or PDD | 1 year
  Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), will combine these tests in order to investigate for their ability to predict successfully whether patients suffered from PDD or DLB.
Symbol digit written predictive for DLB or PDD | 1 year
  Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), will combine these tests in order to investigate for their ability to predict successfully whether patients suffered from PDD or DLB.
Wechsler adult intelligence scale,predictive for DLB or PDD | 1 year
  Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), will combine these tests in order to investigate for their ability to predict successfully whether patients suffered from PDD or DLB.
trail making A and B predictive for DLB or PDD | 1 year
  Two classification algorithms, logistic regression and K-Nearest Neighbors (K-NNs), will combine these tests in order to investigate for their ability to predict successfully whether patients suffered from PDD or DLB.

CONTACTS AND LOCATIONS:
Overall Officials: ANASTASIA BOUGEA, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Anastasia Bougea, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bougea A, Efthymiopoulou E, Spanou I, Zikos P. A Novel Machine Learning Algorithm Predicts Dementia With Lewy Bodies Versus Parkinson's Disease Dementia Based on Clinical and Neuropsychological Scores. J Geriatr Psychiatry Neurol. 2022 May;35(3):317-320. doi: 10.1177/0891988721993556. Epub 2021 Feb 8. PMID 33550890